CLINICAL TRIAL: NCT01462773
Title: A Phase I Study of PS-341 (Bortezomib, Velcade) and Interferon-alpha-2b in Malignant Melanoma.
Brief Title: Study of Patients With Stage IV Malignant Melanoma Using PS-341 (Bortezomib, Velcade) and Interferon-alpha-2b in Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, William Carson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-04105; NCI-2011-03174 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2011-10-19; First posted 2011-10-31 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Melanoma
Keywords: malignant; melanoma
MeSH Terms: conditions — Melanoma | interventions — Bortezomib; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor, interferon therapy) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 8, 15, and 22 and recombinant interferon alfa-2b SC on days 1, 3, and 5 (days 1 and 3 only in week 4 course 1) of weeks 1-4. Treatment repeats every 5 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Bortezomib — VELCADE (1.0 mg/m2, 1.3 mg/m2, or 1.6 mg/m2 IV based on patient cohort). After three patients have received 5 weeks of therapy (1 cycle) at the initial dose of VELCADE (1.0 mg/m2, Cohort 1) with no dose limiting toxicity, the dose will be raised to 1.3 mg/m2 for the next cohort of three patients. If this dose level is well-tolerated in three consecutive patients, the dose of VELCADE will be raised to 1.6 mg/m2.
  Other Names: VELCADE®
Drug: Interferon Alfa-2b — I = IFN-α-2b (INTRON A): 5 million units (MU)/m2 SC. INTRON A (5MU/m2) will be administered subcutaneously on Days 1, 3 and 5 of Week 0. During Cycle I, INTRON A will be administered on Days 1, 3 and 5 of Weeks 1-3 of and on Days 1 and 3 of Week 4 to allow for surgical biopsy on Day 5. During Cycles II-V, IFN-α will be administered on Days 1, 3 and 5 of Weeks 1-4. To assess the toxicity profile of IFN-α-2b alone, no VELCADE will be administered during Week 0.
  Other Names: IFN-α-2b

SUMMARY:
The purpose of this study is to determine the safety, tolerability and dose limiting toxicities (DLTs) of VELCADE when administered in combination with interferon-alpha-2b (IFN-α-2b) to patients with metastatic malignant melanoma.

DETAILED DESCRIPTION:
The primary objective of this study is to:

• Determine the safety, tolerability and DLTs of VELCADE when administered in combination with interferon-alpha-2b (IFN-α-2b) to patients with metastatic malignant melanoma.

The secondary objectives of this study are to:

* Document any objective anti-tumor responses that may occur in response to this treatment regimen.
* Document the time to tumor progression in patients receiving this treatment regimen.
* Measure levels of the cell cycle proteins p21 and p27 in PBMCs and tumor biopsies obtained pre-study and during week 4 of Cycle 1 (Day 26).
* Conduct histologic evaluations of microvessel density, tumor apoptosis and lymphocytic infiltrates within tumor biopsies obtained pre- and post-study.
* Measure plasma levels of bFGF and VEGF over the course of the study.
* Monitor the effects of proteasome inhibition on the biological activity of IFN-α within immune cells by measuring Jak-STAT signal transduction in patient PBMCs.

ELIGIBILITY:
Inclusion Criteria:

* must have histological or cytological diagnosis of cutaneous melanoma and clinical evidence of metastatic, non-resectable regional lymphatic, or extensive in transit recurrent disease. Patients who have had resected metastases will also be eligible provided they have measurable disease.
* have measurable disease. Measurable disease is defined as the presence of at least one measurable lesion.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%).
* Female subjects must be either surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subjects must agree to use an acceptable method for contraception for the duration of the study.
* Patients must have normal organ and marrow function.
* Prior Therapy: Patients with an ECOG performance status of ≤ 2 will be eligible for this protocol regardless of the number of prior treatments provided they have recovered from the reversible effects of prior therapy. Patients are permitted to have received therapy with adjuvant IFN-α2b, if it was completed > 6 months prior to enrollment in the current study.
* Patients with brain metastases are eligible for entry into the study, but must have received definitive therapy consisting of external beam radiation therapy, gamma knife therapy or surgical resection and be clinically stable. Four weeks after the definitive therapy is completed, repeat MRI or CT scans must demonstrate stabilization of disease, and there must be no requirement for Decadron. If the patient does not have brain metastases, then only one brain CT or MRI is required prior to enrollment on study.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

  * Patient has a platelet count of < 100 × 109/L within 14 days before enrollment.
  * Patient has an absolute neutrophil count of < 1.0 x 109/L within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of < 30 mL/minute within 14 days before enrollment.
* Patient has history of significant brain metastases or other clinically significant central nervous system disease.
* Patient has ≥Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patients with evidence of proteinuria on urinalysis.
* Female subject is pregnant or breast-feeding.
* Received other investigational drugs with 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* History of serious psychiatric illness that might be exacerbated by IFN-α-2b.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2010-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Markowitz J, Luedke EA, Grignol VP, Hade EM, Paul BK, Mundy-Bosse BL, Brooks TR, Dao TV, Kondalasula SV, Lesinski GB, Olencki T, Kendra KL, Carson WE 3rd. A phase I trial of bortezomib and interferon-alpha-2b in metastatic melanoma. J Immunother. 2014 Jan;37(1):55-62. doi: 10.1097/CJI.0000000000000009. PMID 24316557
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib & Interferon-a: Bortezomib was administered intravenously weekly along with IFN-a thrice weekly.
Period: Overall Study
Arm/Group | Bortezomib & Interferon-a
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor, Interferon Therapy)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: patients]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Determine Dose Limiting Toxicities (DLTs) of VELCADE When Administered in Combination With IFN-α-2b to Patients With Metastatic Malignant Melanoma.
Description: A standard method for the design of this study. Initially, three patients will be treated at a starting dose of VELCADE (1.0 mg/m2). If one of the three patients demonstrates a DLT, then an additional 3 patients will be treated at that dose level. If only one of the six show DLT, then the next cohort of three patients will be entered at the next dose level (1.3 mg/m2). If two or more of the six demonstrate DLT, no further patients will be treated at that dose level. The highest dose level at which less than 2 patients experienced DLT will be expanded to six patients.
Time Frame: up to 25 weeks or until disease progression
Measure: Number; unit: toxicities
Groups:
- Bortezomib & Interferon-a: Patients were treated on a 5-week cycle. Week 1 of cycle 1, patients received 5 million U/m(2) IFN-a subcutaneously thrice weekly. Weeks 2-4 of cycle 1, bortezomib was administered intravenously weely along with IFN-a thrice weekly. A break from treatment during week 5. Folllowing cycle 1, bortezomib was administered in combination iwth IFN-a. Bortezomib was administered in escalating doses to cohorts of 3 patients.
Arm/Group | Bortezomib & Interferon-a
Number analyzed (Participants) | 16
toxicities
  Grade 4 fatigue | 3
  Grade 4 Lymphopenia | 1

2. Secondary Outcome: Document Any Objective Anti-tumor Responses and Time to Tumor Progression That May Occur in Response to This Treatment Regimen.
Description: * Measure levels of the cell cycle proteins p21 and p27 in PBMCs and tumor biopsies obtained pre-study and during week 4 of Cycle 1 (Day 26).
  * Conduct histologic evaluations of microvessel density, tumor apoptosis and lymphocytic infiltrates within tumor biopsies obtained pre- and post-study.
  * Measure plasma levels of bFGF and VEGF over the course of the study.
  * Monitor the effects of proteasome inhibition on the biological activity of IFN-α within immune cells by measuring Jak-STAT signal transduction in patient PBMCs.
Time Frame: up to 25 weeks
Measure: Number; unit: patients
Arm/Group | Bortezomib & Interferon-a
Number analyzed (Participants) | 16
patients
  partial response | 1
  stable disease | 7

ADVERSE EVENTS:
Description: Adverse events were determined using the NCI CTCAE (Common Terminology Criteria for Adverse Events) version 3.0 as a guideline.
Groups:
- Treatment (Enzyme Inhibitor, Interferon Therapy): Patients were treated on a 5-week cycle. In week 1 of cycle 1, patients received 5 million U/m(2) IFN-α subcutaneously thrice weekly. During weeks 2-4 of cycle 1, bortezomib was administered intravenously weekly along with IFN-α thrice weekly. There was a treatment break during week 5. After cycle 1, bortezomib was administered in combination with IFN-α. Bortezomib was administered in escalating doses (1.0, 1.3, or 1.6 mg/m) to cohorts of 3 patients.
Arm/Group | Treatment (Enzyme Inhibitor, Interferon Therapy)
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Interferon Therapy) (N=16)
Fatigue (General disorders) | 8 (8)
Lymphopenia (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes